CLINICAL TRIAL: NCT03610113
Title: Reverse Shoulder Arthroplasty Versus Conservative Treatment For Complex Proximal Fractures in Elderly Patients
Brief Title: Reverse Or Nothing For Complex Proximal Humeral Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Anoia (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Joan Miquel, Orthopaedic Surgeon, Principal Investigator, Consorci Sanitari de l'Anoia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC12-045
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Humeral Fractures
Keywords: Conservative treatment; Reverse shoulder arthroplasty; Proximal humeral fractures
MeSH Terms: conditions — Humeral Fractures; Shoulder Fractures | interventions — Shoulder Prosthesis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONSERVATIVE TREATMENT (No Intervention): Conservative treatment is conceived to the use of sling for three weeks, followed by rehabilitation protocol
- REVERSE ARTHROPLASTY TREATMENT (Experimental): This group receives a surgical intervention by the use of reverse shoulder arthroplasty through deltopectoral approach and tuberosities reattachment.
  It is followed by the same rehabilitation protocol than conservative treatment
  Interventions: Device: Reverse shoulder arthroplasty

INTERVENTIONS:
Device: Reverse shoulder arthroplasty — The implantation of reverse shoulder prosthesis, and reattachment of greater and lesser tuberosities
  Other Names: Shoulder prosthesis
  Arms: REVERSE ARTHROPLASTY TREATMENT

SUMMARY:
Reverse shoulder prosthesis has recently emerged as an acute treatment for complex proximal humeral fractures. Promising functional results have been reported in observational papers.

However, no clinical trials have yet been reported when comparing the conservative treatment to surgical treatment through the use of reverse shoulder arthroplasty.

DETAILED DESCRIPTION:
Introduction The proximal humeral fractures are frequent in the investigator's environment. Among them, about 20% are considered as complex features. Conservative treatment has traditionally offered an extensive range of results. The reverse shoulder prosthesis as a treatment for acute fractures of the proximal humeral in the elderly population has changed the therapeutic approach of this acute pathology. However, high-level evidence-based studies are still not available, when comparing the conservative treatment with the treatment with reverse shoulder prosthesis.

Objective To compare the functional results and complications of elderly patients presenting acute complex fractures of the proximal humerus through two types of treatments; conservative treatment and treatment with reverse shoulder prosthesis.

Methodology A prospective, multicentre and randomized study comparing conservative treatment with the surgical treatment at two years followup by the use of functional shoulder assessment (Constant scale), complications and re-interventions associated with each treatment. The quality of life will also be analyzed through the SF-36 health questionnaire

Expected results The null hypothesis of the work is based on the appearance of non-significant differences between the two groups of the study (conservative vs. surgical treatment), concerning functional status, complications, and re-interventions

ELIGIBILITY:
Inclusion Criteria:

* Patients with mental conditions available for rehabilitation protocols
* Patients presenting a 3 or 4 part proximal humeral fracture

Exclusion Criteria:

* Extremely displaced fractures with no bony contact or less than 1 cm.
* Cognitive impairment (Pfeiffer test >3)
* Shoulder dislocations
* Unable to sign informed consent or unable to respond to questionnaires
* Trauma or previous surgery of the extremity
* Open or pathological fracture
* Vascular or neurological injury associated
* Unable to collaborate with rehabilitation
* Patients with serious comorbidities that discourage surgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Pain, Mobility, Strenght and Daily Life Activities. (Functional Outcome) | 1 year
  Constant-Murley Score. The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury and it ranges from 0 to 100 points. The test is divided into four subscales: pain (0 to 15 points), activities of daily living (0 to 20 points), strength (0 to 25 points) and range of motion: forward elevation (0 to 10 points), external rotation (o to 10 points), abduction (0 to 10 points) and internal rotation of the shoulder (0 to 10 points). Then, those range of motion items allocate from 0 to 40 points to the global score.
  The higher the score, the higher the quality of the function.

SECONDARY OUTCOMES:
Number of participants with treatment-related surgical reinterventions | 1 year
  Number of participants with treatment-related adverse events that require an additional surgical treatment after the randomization; such as debridement, implant replacement In the control group; reinterventions will be measured by the necessity to receive a treatment for fracture sequelae such as an implantation of a shoulder prosthesis or any other surgical intervention
Number of participants with treatment-related shoulder joint infection | 1 year
  Acute infection will be defined as swelling, erythema, fever, purulent discharge or increasing level of biological parameters such as C-reactive protein (CRP), white blood cell count (WBC).
  Only expected in experimental/intervention group
Number of participants with treatment-related Implant dislocation | 1 year
  It is defined as the number of patients in experimental arm presenting a radiological disalignement between the humeral component (stem) and the glenoid component (glenosphere).
  Only expected in experimental/intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Torrens, PhD, Study Director — Parc de Salut Mar
Locations (1):
- Joan Miquel Noguera, Collbató, Barcelona, Spain

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196